CLINICAL TRIAL: NCT03958123
Title: Evaluation of the Effects of Multiple Therapeutic and Supratherapeutic Doses of Cebranopadol on Cardiac Repolarization in Healthy Subjects
Brief Title: Evaluation of the Effects of Multiple Doses of Cebranopadol on the Electrical Activity of the Heart in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRT-PK-12
Record Dates: First submitted 2019-05-20; First posted 2019-05-21 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Prolonged QTc Interval; Pharmacokinetic
Keywords: QT/QTc Interval
MeSH Terms: interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Participants were randomized to 1 of 4 treatment groups on Day -3: The study included a nested cross-over design for participants in treatment group 3 (A, B).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Group 1: Cebranopadol (Experimental): Supratherapeutic dose (1600 μg) of cebranopadol:
  Participants received placebo once a day for 2 days (Days -3 and -1); 200 μg of cebranopadol once a day for 3 days; 400 μg once a day for 3 days; 600 μg once a day for 3 days; 900 μg once a day for 3 days; 1300 μg once a day for 3 days; 1600 μg once a day for 14 days; and placebo once a day on the last dosing day.
  Participants received capsules under fasting conditions on Days -3, -1, 1, 29 and 30, and under fed conditions on all other dosing days. Participants received four encapsulated cebranopadol/ placebo tablets and 1 encapsulated moxifloxacin/ placebo tablet (5 capsules in total) on Day -3, Day -1, and from Day 1 to Day 30. Capsules were taken with 240 mL of water.
  Interventions: Drug: 100 μg cebranopadol; Drug: 200 μg cebranopadol; Drug: 400 μg cebranopadol; Drug: Placebo to cebranopadol encapsulated tablets; Drug: Placebo to moxifloxacin encapsulated tablets
- Treatment Group 2: Cebranopadol (Experimental): Therapeutic dose (600 μg) of cebranopadol:
  Participants received placebo once a day for the first 11 days (Days -3, -1 and 1-9); 200 μg of cebranopadol once a day for 3 days; 400 μg once a day for 3 days; 600 μg once a day for 14 days; and placebo once a day on the last dosing day.
  Participants received capsules under fasting conditions on Days -3, -1, 1, 29 and 30, and under fed conditions on all other dosing days. Participants received 4 encapsulated cebranopadol/ placebo tablets and 1 encapsulated moxifloxacin/ placebo tablet (5 capsules in total) on Day -3, Day -1, and from Day 1 to Day 30. Capsules were taken with 240 mL of water.
  Interventions: Drug: 200 μg cebranopadol; Drug: 400 μg cebranopadol; Drug: Placebo to cebranopadol encapsulated tablets; Drug: Placebo to moxifloxacin encapsulated tablets
- Treatment Group 3A: Placebo and Moxifloxacin (Experimental): Placebo / Moxifloxacin:
  Participants received placebo once a day for 31 days (Days -3, -1 and 1-29) and moxifloxacin 400 mg once on the last dosing day. Participants received capsules under fasting conditions on Days -3, -1, 1, 29 and 30, and under fed conditions on all other dosing days.
  Participants received 4 encapsulated cebranopadol/ placebo tablets and 1 encapsulated moxifloxacin/ placebo tablet (5 capsules in total) on Day -3, Day -1, and from Day 1 to Day 30. Capsules were taken with 240 mL of water.
  Interventions: Drug: Placebo to cebranopadol encapsulated tablets; Drug: 400 mg Moxifloxacin; Drug: Placebo to moxifloxacin encapsulated tablets
- Treatment Group 3B: Moxifloxacin and Placebo (Experimental): Moxifloxacin / Placebo:
  Participants received placebo once a day for 2 days (Days -3 and -1); moxifloxacin 400 mg once for 1 day; and placebo once a day for the following 29 days. Participants received capsules under fasting conditions on Days -3, -1, 1, 29 and 30, and under fed conditions on all other dosing days.
  Participants received four encapsulated cebranopadol/ placebo tablets and 1 encapsulated moxifloxacin/ placebo tablet (5 capsules in total) on Day -3, Day -1, and from Day 1 to Day 30. Capsules were taken with 240 mL of water.
  Interventions: Drug: Placebo to cebranopadol encapsulated tablets; Drug: 400 mg Moxifloxacin; Drug: Placebo to moxifloxacin encapsulated tablets

INTERVENTIONS:
Drug: 100 μg cebranopadol — Encapsulated 100 μg cebranopadol tablet.
  Arms: Treatment Group 1: Cebranopadol
Drug: 200 μg cebranopadol — Encapsulated 200 μg cebranopadol tablet.
  Arms: Treatment Group 1: Cebranopadol; Treatment Group 2: Cebranopadol
Drug: 400 μg cebranopadol — Encapsulated 400 μg cebranopadol tablet.
  Arms: Treatment Group 1: Cebranopadol; Treatment Group 2: Cebranopadol
Drug: Placebo to cebranopadol encapsulated tablets — Matching placebo to cebranopadol encapsulated tablet.
Drug: 400 mg Moxifloxacin — Encapsulated 400 mg moxifloxacin tablet.
  Arms: Treatment Group 3A: Placebo and Moxifloxacin; Treatment Group 3B: Moxifloxacin and Placebo
Drug: Placebo to moxifloxacin encapsulated tablets — Matching placebo to moxifloxacin (400 mg) encapsulated tablet.

SUMMARY:
The objective of this study was to evaluate the effects of cebranopadol (GRT6005) on the electrical activity of the heart in healthy participants.

The study consisted of a screening period within 21 days before the first dose of investigational medicinal product (IMP) (between Day -25 and Day -4) during which informed consent was obtained and the general suitability of the participants for the trial was assessed according to the inclusion/exclusion criteria.

Participants were confined to the trial site from 4 days before first IMP dosing on Day 1 to 4 days after last IMP dosing on Day 30. During this period, multiple-doses of cebranopadol or matching placebo and a single-dose of moxifloxacin or matching placebo were administered. Moxifloxacin was used as a positive control. It has consistently shown that it has an effect on the heart rhythm. Continuous 12-lead ECGs were recorded at defined time points. Multiple blood and urine samples were drawn for pharmacokinetic evaluations and safety laboratory monitoring (hematology, chemistry, and urinalysis). Additional safety evaluations included recording of adverse events, vital signs (systolic and diastolic blood pressure, pulse rate, respiration rate, body temperature, and weight), oxygen saturation, standard 12-lead ECG, Clinical Opiate Withdrawal Scale (COWS) assessment, and Columbia-Suicide Severity Rating Scale (C-SSRS) assessment.

An End-of-Trial Visit was performed on Day 34, or within 7 days after the last pharmacokinetic sample on Day 34, or at early withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form (ICF) and have the mental capability to understand it.
* Be a healthy male or female, aged 18 through 45 years, inclusive.
* If female, have a negative result from a serum pregnancy test at screening and a negative result from a serum or urine pregnancy test on Day -4.
* If male, agree to use an effective method of contraception (ie, condom plus diaphragm with spermicide or condom plus spermicide) and not have their partners become pregnant throughout the study, or have been sterilized for at least 1 year (with supporting documentation of the absence of sperm in the ejaculate postvasectomy).
* If female of childbearing potential, agree to use an effective method of contraception (ie, condom plus diaphragm with spermicide, condom plus spermicide, or nonhormonal intrauterine device) and not become pregnant throughout the study. Females who are at least 2-years postmenopausal (with supporting documentation from an obstetrician/gynecologist) or who have had tubal ligation or hysterectomy (with supporting documentation from the physician who performed the surgery) will not be considered to be of childbearing potential.
* Be nonsmoking (never smoked or have not smoked within the previous 2 years).
* Have a body mass index (BMI) greater than or equal to 18 kilograms per square meter and less than or equal to 30 kilograms per square meter.
* Have a sitting pulse rate greater than or equal to 50 beats per minute (bpm) and less than or equal to 100 bpm during the vital sign assessment at screening.

Exclusion Criteria:

* Known hypersensitivity to cebranopadol, other opioids, or moxifloxacin or other fluoroquinolone antibiotics.
* Clinically significant disease state, in the opinion of the examining physician, in any body system.
* Sitting systolic blood pressure (BP) greater than or equal to 140 millimeters mercury (mm Hg) or less than or equal to 90 mm Hg or sitting diastolic BP greater than or equal to 90 mm Hg or less than or equal to 50 mm Hg at screening.
* Abnormal electrocardiogram (ECG) results thought to be potentially clinically significant (PCS), or QT prolongation (QTcF greater than or equal to 450 milliseconds (msec) or uncorrected QT greater than or equal to 500 msec) according to the Investigator.
* History of cardiovascular disease including but not limited to long QT syndrome (or family history of long QT syndrome), cardiac arrhythmia, orthostatic hypotension, and coronary artery or valvular disease.
* Positive test results for anti-human immunodeficiency virus type 1, hepatitis B surface antigen, hepatitis B core antibodies, or anti-hepatitis C virus at screening.
* Abnormal and clinically significant results on medical history, physical examination, serum chemistry, hematology, or urinalysis.
* History of alcohol or other substance abuse within the previous 5 years.
* Positive urine drug screen test results for benzoylecgonine (cocaine), methadone, barbiturates, amphetamines, benzodiazepines, alcohol, cannabinoids, opiates, phencyclidine, or cotinine at screening or Day -4.
* Have taken opioids within the past 1 month.
* Participation in any other clinical investigation using an experimental drug requiring repeated blood or plasma draws within 60 days of investigational product administration.
* Participation in a blood or plasma donation program within 60 or 30 days, respectively, of investigational product administration.
* Consumption of caffeine products within 48 hours or any grapefruit-containing products or Seville oranges within 14 days or consumption of alcohol or poppy seeds within 72 hours before administration of investigational product.
* Consumption of beverages or food containing quinine (bitter lemon, tonic water) within 14 days before administration of investigational product until discharge from the study center.
* Have any clinical condition that might affect the absorption, distribution, biotransformation, or excretion of cebranopadol or moxifloxacin.
* Employee, or immediate relative of an employee, of Forest Laboratories, Inc. or Grünenthal GmbH, any of its affiliates or partners, or the study center.
* Taken any concomitant medications (including over-the-counter medications) within 14 days or hormonal drug products within 30 days before administration of investigational product.
* Previously taken cebranopadol or previously participated in an investigational study of cebranopadol.
* Breastfeeding.
* Responses to the Columbia-Suicide Severity Rating Scale (C-SSRS) that indicate any current suicidal ideation or a history of active suicidal ideation or suicide attempts.
* Suicidal risk based on the opinion of the principal investigator (or appropriately trained designee).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2013-11-27 (Actual); Study Completion 2013-11-27 (Actual)

PRIMARY OUTCOMES:
QTcNi change from time-matched baseline measurement on Day -1 to Day 29 - supported sitting position | Day -1 up to Day 29
  Largest time-matched mean difference between cebranopadol and placebo in supported sitting QT interval corrected for heart rate using an individual correction (QTcNi) change from time-matched baseline measurement on Day -1.

SECONDARY OUTCOMES:
QTcNi change from time-matched baseline measurement on Day -1 to Day 29 - supine position | Day -1 up to Day 29
  Largest time-matched mean difference between cebranopadol and placebo in supine QTcNi change from time-matched baseline measurement on Day -1.
QTcF change from time-matched baseline measurement on Day -1 to Day 29 - sitting position | Day -1 up to Day 29
  Largest time-matched mean difference between cebranopadol and placebo in supported sitting QT interval corrected for heart rate using the Fridericia formula (QTcF) change from time-matched baseline measurement on Day -1.
QTcF change from time-matched baseline measurement on Day -1 to Day 29 - supine position | Day -1 up to Day 29
  Largest time-matched mean difference between cebranopadol and placebo in supine QTcF change from time-matched baseline measurement on Day -1.
Pharmacokinetic parameter: AUC0-tau,ss of cebranopadol | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to the end of the dosing interval, tau, at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-tau,ss of M2 (7-hydroxy-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to the end of the dosing interval, tau, at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-tau,ss of M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to the end of the dosing interval, tau, at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-tau,ss of M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to the end of the dosing interval, tau, at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-t of cebranopadol | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to time t after the last dose. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-t of M2 (7-hydroxy-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to time t after the last dose. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-t of M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to time t after the last dose. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-t of M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to time t after the last dose. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cav,ss of cebranopadol | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Average plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cav,ss of M2 (7-hydroxy-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Average plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cav,ss of M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Average plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cav,ss of M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Average plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmax,ss of cebranopadol | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Maximum plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmax,ss of M2 (7-hydroxy-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Maximum plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmax,ss of M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Maximum plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmax,ss of M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Maximum plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmin,ss of cebranopadol | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Minimum plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmin,ss of M2 (7-hydroxy-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Minimum plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmin,ss of M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Minimum plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmin,ss of M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Minimum plasma drug concentration at steady state. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Fluctuation of cebranopadol | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  The difference between Cmin and Cmax standardized to Cavg, within 1 dosing interval. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Fluctuation of M2 (7-hydroxy-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  The difference between Cmin and Cmax standardized to Cavg, within 1 dosing interval. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Fluctuation of M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  The difference between Cmin and Cmax standardized to Cavg, within 1 dosing interval. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Fluctuation of M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  The difference between Cmin and Cmax standardized to Cavg, within 1 dosing interval. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Swing of cebranopadol | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  The difference between Cmin and Cmax standardized to Cmin, within 1 dosing interval. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Swing of M2 (7-hydroxy-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  The difference between Cmin and Cmax standardized to Cmin, within 1 dosing interval. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Swing of M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  The difference between Cmin and Cmax standardized to Cmin, within 1 dosing interval. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Swing of M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  The difference between Cmin and Cmax standardized to Cmin, within 1 dosing interval. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: tmax of cebranopadol | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Time of maximum plasma drug concentration. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: tmax of M2 (7-hydroxy-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Time of maximum plasma drug concentration. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: tmax of M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Time of maximum plasma drug concentration. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: tmax of M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Time of maximum plasma drug concentration. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-inf of moxifloxacin | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the plasma concentration versus time curve from time 0 to infinity. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for moxifloxacin were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: AUC0-t of moxifloxacin | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Area under the first moment of the plasma concentration versus time curve from time 0 to time t. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for moxifloxacin were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: Cmax of moxifloxacin | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Maximum plasma drug concentration. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for moxifloxacin were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: t1/2 of moxifloxacin | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Terminal half-life. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for moxifloxacin were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.
Pharmacokinetic parameter: tmax of moxifloxacin | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 14, 24, 48, 72, and 96 hours post-dose
  Time of maximum plasma drug concentration. PK blood samples were collected before administration of the IMP and up to 96 hours after dosing; 32 PK blood samples were obtained from each participant. Plasma concentrations for moxifloxacin were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Grünenthal, Study Director — Grünenthal GmbH
Locations (1):
- US001 Contract research organization, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No